CLINICAL TRIAL: NCT00026962
Title: Assessment of the Effects of Raloxifene on Salivary Estradiol and Progesterone Levels
Brief Title: Effects of Raloxifene on Hormone Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990180; 99-C-0180
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-08

CONDITIONS: Breast Cancer
Keywords: Breast; Hormones; Prevention; Saliva; Serum
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: measuring estradiol and progesterone levels in saliva

SUMMARY:
Blood levels of the hormones estradiol and progesterone are of interest in evaluating ovarian function. However, because these hormone levels vary from day to day, blood samples must be taken very often or elaborately timed to specific phases of the menstrual cycle. A method has now been developed for measuring estradiol and progesterone levels in saliva. This study will test the accuracy of this method and examine whether salivary levels of these hormones change after treatment with raloxifene.

Hormone levels will be measured during 3 menstrual cycles in women currently enrolled in the clinical study, "A Phase II Trial of Two Doses of Raloxifene in Women at Risk of Developing Invasive Breast Cancer." Participants will provide a saliva sample every morning for about a month during three collection periods-1 month before beginning raloxifene treatment, and 3 and 12 months after treatment starts. Patients will be given kits for collecting the samples and mailing them to the laboratory at the end of each collection period.

DETAILED DESCRIPTION:
Deviations from normal levels of serum E(2) and P are of interest in evaluating ovarian function. However, the day-to-day variations in these levels necessitates serial blood sampling or elaborate efforts to time blood draws within specific phases of the menstrual cycle. A noninvasive method for assessment of the levels of sex steroids on a daily basis using saliva has been developed. This study will assess the levels of estradiol and progesterone during 3 menstrual cycles (pre-drug and after 3 and 12 months of raloxifene therapy) in pre-menopausal women participating in a pilot chemoprevention trial of raloxifene.

ELIGIBILITY:
Patients must be enrolled on protocol 98-C-0123 (MB #402) or this same protocol at the National Naval Medical Center.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1999-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Read GF. Status report on measurement of salivary estrogens and androgens. Ann N Y Acad Sci. 1993 Sep 20;694:146-60. doi: 10.1111/j.1749-6632.1993.tb18349.x. No abstract available. PMID 8215051
- [Background] Rosner W. The functions of corticosteroid-binding globulin and sex hormone-binding globulin: recent advances. Endocr Rev. 1990 Feb;11(1):80-91. doi: 10.1210/edrv-11-1-80. No abstract available. PMID 2180689
- [Background] Petra PH. The plasma sex steroid binding protein (SBP or SHBG). A critical review of recent developments on the structure, molecular biology and function. J Steroid Biochem Mol Biol. 1991;40(4-6):735-53. doi: 10.1016/0960-0760(91)90299-k. PMID 1958572